CLINICAL TRIAL: NCT03452241
Title: Long-term Follow-up Study of Substance Abuse Screening and Intervention in Multi Primary Care Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, DU, Jiang, Principal Investigator, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: JDu-004
Record Dates: First submitted 2018-01-19; First posted 2018-03-02 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Substance Use
Keywords: Screening, Brief Intervention, and Referral to Treatment; Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group (Experimental): The medical staffs who received the training will use the manual of brief intervention to deliver it and other materials about the harm of substance use.
  Interventions: Other: Intervention Group
- Control Group (Other): The participants only receive the materials about the harm of substance use
  Interventions: Other: Control Group
- Intervention Group 1 (Experimental): The medical staffs who received the training will use the manual of brief intervention twice to deliver it and other materials about the harm of substance use.
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — The medical staffs who received the training will use the manual of brief intervention to deliver BI and other materials about the harm of substance use.BI refers to a standard 15-30 minute intervention that includes a series of standard models that stimulate knowledge, motivation and behavior that reduce substance abuse.the harm of substance use is a dedicated paper publicity handbook, written by the SHMC, detailing the hazards of substance abuse.
  Arms: Intervention Group; Intervention Group 1
Other: Control Group — The participants only receive the materials about the harm of substance use.the harm of substance use is a dedicated paper publicity handbook, written by the SHMC, detailing the hazards of substance abuse.
  Arms: Control Group

SUMMARY:
The purpose of this research is to improve the ability of primary medical staffs in screening and intervention for alcohol, benzodiazepines, and other illicit drug use.

DETAILED DESCRIPTION:
In order to reduce the social and personal harm caused by drugs, it is urgent to strengthen the ability of the primary health institutions in screening and intervention the addictive substances use. Firstly, the investigators will invite 10 primary medical staffs and 10 experts in addition to revise the manual of Alcohol, Smoking, and Substance Use Involvement Screening Test (ASSIST) and Brief Intervention (BI). Then, the investigators will recruit related medical staffs in five provinces to participate the training of ASSIST and BI. Secondly, the researcher will investigate the effects of BI technology in reducing the use of addictive substances, improve the addiction related knowledge of patients through randomized controlled study. Finally, the investigators will collect the research information, revise the manual, and promote the training.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 years;
* the patient to the community medical institutions;
* ASSIST score is in 12-27, in a moderate risk;
* voluntary to participate;
* to agree to complete baseline interviews and follow-up studies

Exclusion Criteria:

* unable to complete the questionnaire;
* serious physical illness, action inconvenience.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2018-04-14 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in risk behaviors at 1 and 3 month | baseline, 1 and 3 month
  Risk Behaviors will be measured by ASSIST questionnaire.

SECONDARY OUTCOMES:
Knowledge related to Substance Use measured by Knowledge related to Addiction questionnaire | baseline, 1 and 3 month
  Knowledge related to substance use will be measured by Knowledge related to Addiction questionnaire
Motivation measured by Pre-treatment Readiness Scale | baseline, 1 and 3 month
  PRSS is a 5-point scale and the highest score at any stage represents the patient at this stage.
Depression measured by Self-Rating Depression Scale (SDS) | baseline, 1 and 3 month
  SDS contains 20 items and the standard total score is 53, 53-62: mild to mild depression; 63-72: moderate to severe;> 72: severe depression
Anxiety measured by Self-Rating Anxiety Scale (SAS). | baseline, 1 and 3 month
  SDS contains 20 items. According to the Chinese norm results, the standard points of the cut-off value is 50 points, of which 50-59 is divided into mild anxiety, 60-69 is divided into moderate anxiety, 70 points for severe anxiety
Self-esteem measured by Self-esteem questionnaire | baseline, 1 and 3 month
  the change of self-esteem will be measured by Self-esteem questionnaire.
Positive and Negative Affect measured by Positive and Negative Affect Scale (PANAS) | baseline, 1 and 3 month
  It contains 20 entries. A high positive emotional score indicates an individual's energy, concentration, and emotional well-being while a low score indicates indifference. Negative emotional high points that the individual subjective feeling puzzled, painful emotional state, while the score is low that calm.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D, Principal Investigator — Study Principal Investigator Shanghai Mental Health Center
Locations (1):
- Henan Provincical Peoples Hospital, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu R, Yuan C, Sun W, Wang W, Zhang L, Zhai J, Guan Q, Wu X, Long J, Zhao M, Du J. Effectiveness of E-SBIRT intervention in community healthcare institution in China: study proposal for a randomised controlled trial. Gen Psychiatr. 2021 Sep 24;34(5):e100486. doi: 10.1136/gpsych-2021-100486. eCollection 2021. PMID 34651102